CLINICAL TRIAL: NCT02952378
Title: Volume Kinetics for Hyperoncotic Albumin in Burn Patients as Well as for Healthy Subjects
Acronym: VAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, Assoc prof, University Hospital, Linkoeping
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAB
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Albumins; galactosamine-conjugated serum albumin-conjugated-(rhodamine X)20

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Burn patients (Experimental): Patients with burns exceeding 6-8 Total Burned Surface Area %
  Interventions: Drug: Albumins
- Healthy individuals (Experimental): Healthy individuals without allergies.
  Interventions: Drug: Albumins

INTERVENTIONS:
Drug: Albumins — Infusion of 3ml/kg bodyweight of hyperoncotic albumin 20% during 30 minutes.
  Other Names: Albumin 20%

SUMMARY:
Treatment with colloidal solutions has during long time been a cornerstone within intensive care. Lately, doubts have been raised about synthetic colloids, and the natural albumin has been used more and more.

One of these solutions is the hyperoncotic "Albumin 20%". However there are still many aspects of the physiological effects of hyperoncotic albumin, that are not known. In this study physiological effects will be studied in burn patients and healthy subjects. The colloid osmotic pressure and the increase of the plasma volume will be measured in 15 healthy subjects and in 15 burn patients. The effect on the plasma volume will be studied using hemoglobin as a marker of dilution. Colloids osmotic pressure and albumin concentration will be measured directly and urin production will also be measured. Blood samples will be collected during 4 to 5 hours to achieve a profile over the changes.

DETAILED DESCRIPTION:
Healthy individuals are asked to refrain from eating and drinking the night before the study. Two hours before study start, the subjects may take a sandwich and a glas to drink. Patients will also be asked to keep the same rules unless they receive parenteral nutrition. Shortly before the study, the subjects are asked to leave an urine sample.

After 15 minutes of rest the first bood samples are taken. An infusion 3 ml/kg bodyweight Albumin 20% is given during 30 minutes. The first hour after study start (start of infusion) blood samples are taken every 10 minutes. The following 4 hours another 9 blood samples are collected. Hemoglobin, albumin and colloidosmotic pressure will be measured at every occasion.

C-reactive protein, interleukin-6, Syndecan -1 as well as heparan sulfate, will be measured before, after 1 hour and 5 hours after study start.

The total volume of blood collected will be 150 ml. If the study subjects have a low urin output, acetated Ringers will be given at the end of the study. Liberal fluid intake is recommended the same day and the next.

ELIGIBILITY:
Inclusion Criteria:

* For healthy individuals: Healthy, without allergies and with the age of 18 years or above.
* For patients: Burn injury exceeding 6-8 Total Burned Surface Area %

Exclusion Criteria:

* Heart failure
* Signs of kidney injury/failure
* Severe allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma volume | 5 hours
  Plasma volume expansion using hemoglobin as a marker of dilution.

SECONDARY OUTCOMES:
Colloid osmotic pressure | 5 hours
  Effect of hyperoncotic albumin on oncotic pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Zdolsek, MD,PhD,Assoc prof, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- Burn ward, University Hospital, Linköping, Linköping, Sweden

REFERENCES:
- [Derived] Hahn RG, Zdolsek M, Krizhanovskii C, Ntika S, Zdolsek J. Elevated Plasma Concentrations of Syndecan-1 Do Not Correlate With Increased Capillary Leakage of 20% Albumin. Anesth Analg. 2021 Mar 1;132(3):856-865. doi: 10.1213/ANE.0000000000005315. PMID 33350618
- [Derived] Zdolsek M, Hahn RG, Sjoberg F, Zdolsek JH. Plasma volume expansion and capillary leakage of 20% albumin in burned patients and volunteers. Crit Care. 2020 May 5;24(1):191. doi: 10.1186/s13054-020-02855-0. PMID 32366324